CLINICAL TRIAL: NCT00178711
Title: National Acute Brain Injury Study: Hypothermia IIR
Brief Title: Effects of Hypothermia Upon Outcomes After Acute Traumatic Brain Injury
Acronym: NABIS:HIIR
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Futility
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Guy Clifton, Professor - Neurosurgery, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5U01NS043353-06 (NIH); FDA-2014-109 (Other: FDA)
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Results first posted 2014-08-11 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; Hypothermia
MeSH Terms: conditions — Brain Injuries, Traumatic; Hypothermia | interventions — Hypothermia, Induced

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hypothermia (Active Comparator): Induction and maintenance of moderate hypothermia to 33 degrees celsius achieved within 2.5 hours of injury and maintained for 48 hours.
  Interventions: Device: Hypothermia
- control (No Intervention): treated at normothermia

INTERVENTIONS:
Device: Hypothermia — Induction of moderate hypothermia to 33 degrees celsius, within 2.5 hours from time of injury and maintained for 48 hours
  Other Names: moderate hypothermia
  Arms: hypothermia

SUMMARY:
Induction of hypothermia to < 35˚C by < 2.5 hours after severe traumatic brain injury, reaching 33˚C by 4 hours after injury and maintained for 48 hours in patients aged 16-45 will result in an increased number of patients with good outcomes at six months after injury compared to patients randomized to normothermia.

DETAILED DESCRIPTION:
NABIS:HIIR was a randomized clinical trial conducted in patients with severe brain injury, age 16-45. Patients were randomized to standard treatment at normothermia or to standard treatment with moderate hypothermia (32.5-34C for 48 hours). An intent to treat analysis was used with the primary outcome measure as the Glasgow Outcome Scale at six months after injury. GOS is dichotomized into good outcome (Good Recovery/Moderate Disability) and poor outcome (Severe Disability, Vegetative, Dead).

ELIGIBILITY:
Inclusion Criteria:

1. Non-penetrating brain injury with post-resuscitation Glasgow Coma Score (GCS) < 8 (motor 1-5)
2. Estimated or known age > 16 and < 45 years old
3. Time of Injury within 2.5hrs of arrival at hospital

Exclusion Criteria:

1. GCS = 7 or 8 with a normal head Cat Scan (CT) scan or showing only mild Subarachnoid hemorrhage (SAH)or skull fracture or GCS > 9 post- randomization
2. GCS = 3 AND bilaterally non-reactive pupils
3. Abbreviated Injury Score (AIS) > 4 for any body area except head
4. Positive abdominal ultrasound or CT scan
5. Persistent hypotension (systolic blood pressure < 110mmHGg)
6. Persistent hypoxia (O2 Saturation < 94%)
7. Positive pregnancy test
8. Injured greater than 2.5 hours from hospital arrival
9. Pre-existing medical conditions, if known

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 232 (Actual)
Dates: Start 2005-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guy L Clifton, MD, Principal Investigator — UTHSC-H
Locations (5):
- United States (4):
  - University of St Louis : St. Louis University Hospital, St Louis, Missouri
  - University of Pittsburgh : University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Texas Health Science Center, Memorial Hermann Hospital, Houston, Texas
  - Charleston Area Medical Center, Charleston, West Virginia
- University of Calgary Health Science Center : Foothills Medical Center, Calgary, Alberta, Canada

REFERENCES:
- [Result] Clifton GL, Coffey CS, Fourwinds S, Zygun D, Valadka A, Smith KR Jr, Frisby ML, Bucholz RD, Wilde EA, Levin HS, Okonkwo DO. Early induction of hypothermia for evacuated intracranial hematomas: a post hoc analysis of two clinical trials. J Neurosurg. 2012 Oct;117(4):714-20. doi: 10.3171/2012.6.JNS111690. Epub 2012 Jul 27. PMID 22839656
- [Result] Clifton GL, Valadka A, Zygun D, Coffey CS, Drever P, Fourwinds S, Janis LS, Wilde E, Taylor P, Harshman K, Conley A, Puccio A, Levin HS, McCauley SR, Bucholz RD, Smith KR, Schmidt JH, Scott JN, Yonas H, Okonkwo DO. Very early hypothermia induction in patients with severe brain injury (the National Acute Brain Injury Study: Hypothermia II): a randomised trial. Lancet Neurol. 2011 Feb;10(2):131-9. doi: 10.1016/S1474-4422(10)70300-8. Epub 2010 Dec 17. PMID 21169065

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled in hospitals of University of Texas Health Science Center at Houston, University of Calgary, University of Pittsburgh, St. Louis University, Charleston Area Medical Center, and University of New Mexico.Enrollment occurred from December 2005 to June 2009 with follow-up from June 2006 through December 2009
Pre-assignment Details: Enrollment criteria at the first eligibility assessment were ages 16-45, non-penetrating brain injury, and not responsive to instructions. 232 participants met these criteria and also had none of a first set of exclusion criteria. At the second eligibility assessment, 97 patients had none of a second set of exclusion criteria.
Groups:
- Hypothermia: There were two sets of exclusion criteria-one in the field; the other after resuscitation in the ER. In the field, patients were excluded for suspected pregnancy, systolic blood pressure <110 mm Hg, diastolic blood pressure <60 mm Hg, sustained heart rate >120 beats per minute, or failure to be reached by study-affiliated personnel within 2.5 hours of injury.
  Those that did not have any of the first set of exclusion criteria were further assessed for the presence of Glasgow Coma Scale 3-8 without life-threatening associated injuries. The second set of exclusion criteria were GCS 3 with nonreactive pupils, GCS 7-8 with normal brain CT scan, inability to obtain an accurate GCS, Abbreviated Injury Severity Score >4 for organs other than brain4, systolic blood pressure <110 mm Hg or diastolic blood pressure <60 mm Hg, persistent hypoxia, (oxygen saturation < 94%), or positive pregnancy test.
- Control: 45 patients who had none of the second set of exclusion criteria and who has been randomized to normothermia served as the control group
Period: Overall Study
Arm/Group | Hypothermia | Control
Started | 52 | 45
Completed | 52 | 45
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: hypothermia group-- 26 ± 9 years of age, 40 males/12 females normothermia group--31 ± 11 year of age, 41 males/4 females
Groups:
- Hypothermia: Induction and maintenance of moderate hypothermia to 33 degrees celsius achieved within 4 hours of injury and maintained for 48 hours.
  Hypothermia: Induction of moderate hypothermia to 33 degrees celsius, within 4 hours from time of injury and maintained for 48 hours
- Total: Total of all reporting groups
Arm/Group | Hypothermia | Control | Total
Number analyzed (Participants) | 52 | 45 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (9) | 31 (11) | 28 (10)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 6 | 13
  Between 18 and 65 years | 45 | 38 | 83
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 4 | 16
  Male | 40 | 41 | 81

OUTCOME MEASURES:

1. Primary Outcome: The Dichotomized Glasgow Outcome Scale
Description: The primary outcome measure was the Glasgow Outcome Scale measured in person six months after injury by examiners who were blinded to the patient's treatment group. Good recovery and moderate disability were designated as favorable outcomes; severe disability, a vegetative state, and death as poor outcomes.
Time Frame: 6 months with a window of plus or minus one month
Population: Intention to Treat
Measure: Number; unit: participants with a poor outcome
Arm/Group | Hypothermia | Control
Number analyzed (Participants) | 52 | 45
participants with a poor outcome | 31 [0.76 to 1.53] | 25 [0.76 to 1.53]
Statistical Analysis 1: Comparison: Hypothermia vs Control; The primary hypothesis was a two-sided test assessing whether the induction of hypothermia modified the percentage of subjects with poor outcomes at 6 months after injury. Percentages in each group were compared using a generalized linear model with a binomial distribution and log link function, logistic regression model with admission age and baseline GCS as covariates; Test type: Superiority or Other; p = 0.67, Regression, Logistic; Risk Ratio (RR) = 1.08, 95% CI 2-sided [0.76 to 1.53]

2. Other Pre Specified Outcome: Glasgow Outcome Scale - Extended
Time Frame: 0-12 months
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Disability Rating Scale
Time Frame: assessed 0-12 months
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Neurobehavioral Rating Scale - Revised
Time Frame: 0-12 months
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Neurological Outcome Scale for Traumatic Brain Injury
Time Frame: 0-12 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Symbol Digit Modalities Test
Time Frame: 0-12 months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Rey Osterrieth Complex Figure
Time Frame: 0-12 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Verbal Selective Reminding Test Trails B
Time Frame: 0-12 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Grooved Pegboard
Time Frame: 0-12 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Controlled Oral Word Association Test
Time Frame: 0-12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the time of the second eligibility assessment to the time of discharge from the acute-care hospital. Generally patients were discharged from the acute care hospital within 3 months of admission.
Groups:
- Randomized to Hypothermia and Hypothermia Maintained: Induction and maintenance of moderate hypothermia and not excluded by second set of exclusion criteria
- Randomized to Normothermia and Normothermia Maintained: Induction and maintenance of normothermia and not excluded by second set of exclusion criteria
- Randomized to Hypothermia and Then Excluded: Induction and maintenance of moderate hypothermia before trauma evaluation in ED and then excluded by second set of criteria
- Randomized to Normothermia Then Excluded: Maintenance of normothermia before trauma evaluation in ED and then excluded by second set of criteria
Arm/Group | Randomized to Hypothermia and Hypothermia Maintained | Randomized to Normothermia and Normothermia Maintained | Randomized to Hypothermia and Then Excluded | Randomized to Normothermia Then Excluded
Serious Adverse Events (participants affected / at risk) | 30/52 | 20/45 | 11/67 | 5/68
Other Adverse Events (participants affected / at risk) | 42/52 | 38/45 | 22/67 | 30/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized to Hypothermia and Hypothermia Maintained (N=52) | Randomized to Normothermia and Normothermia Maintained (N=45) | Randomized to Hypothermia and Then Excluded (N=67) | Randomized to Normothermia Then Excluded (N=68)
Elevated Intracranial Pressure (Nervous system disorders) | 14 (91) | 9 (20) | 4 (7) | 0 (0) — Intracranial pressure levels greater than 30mmHg for more than 30 minutes or levels greater than 40 mmHg for 5 minutes, non-responsive to maximal medical management and requires initiation of barbiturate coma.
Decreased Cerebral Perfusion Pressure (Nervous system disorders) | 21 (46) | 13 (34) | 4 (15) | 0 (0) — Cerebral perfusion pressure <50 mmHg for each occurrence documented on the physiology case report form during hourly data collection
Subdural Hemorrhage (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — New hemorrhage into subdural space requiring surgery
Intraparenchymal Hemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — New hemorrhage into brain tissue requiring surgery
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — acute hypoxia associated with high probability ventilation-perfusion scan, positive Spiral CT scan, computed tomography angiography or MRI associated with hypotension or persistent SaO2 less than 90% for greater than or equal to 2 hours
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) — Presence of all 3 of the following; 1. bilateral pulmonary infiltrates 2. a PCWP<18 mm Hg 3. a consistent PO2:FiO2 ratio of <200 for greater than or equal to 3 hours
Hypothermia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — rectal or core temperature less than or equal to 32 degrees C for any period of time not induced or related to general anesthesia
Multiple Organ Dysfunction (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) — a pattern of simultaneous or near simultaneous organ failure in at least 3 organ systems.
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — pO2 <50 mm Hg on greater than or equal to 70% FIO2 or persistent O2 saturation <94% for greater than or equal to 2 hours
Hypotension (Cardiac disorders) | 1 (6) | 0 (0) | 1 (1) | 0 (0) — systolic blood pressure < 90 mm Hg or Mean Arterial Pressure < 70 mm Hg for 2 or more consecutive hours associated with end-organ failure due to hypo-perfusion
Cardiac Arrest (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) — sudden or unexpected cessation of pumping action of the heart
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — presence of blood in the pleural cavity which is not present on admission chest x-ray which drains >200 ml/hr for greater than or equal to 2 hours
Tentorial Herniation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — acute clinical neurologic deterioration with pupillary dilation
Blood Stream Infection (Infections and infestations) | 0 (0) | 2 (2) | 3 (4) | 3 (3) — Has a recognized pathogen from 1 or more blood cultures and organism is not related to infection at another site; or has fever >38C or chills or hypotension and positive blood culture
Catheter Positive Culture (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — >15 colonies of pathogenic microorganisms cultured from an arterial or central venous catheter tip associated with clinical sepsis or laboratory-confirmed bloodstream infection
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Presence of air in the pleural cavity which is not present on admission x-ray associated with hypoxemia or respiratory distress
Epidural Hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — New hemorrhage into epidural space. (Does not include EDH from initial injury but includes a re-bleed into the previously evacuated surgical site
Clinical Sepsis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — At least one of following: fever > 38 degrees C SBP < 90 mmHg oliguria (< 20 cc/hr) AND blood culture NOT done or NO organisms in blood no apparent infection at another site physician institutes treatment for sepsis
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized to Hypothermia and Hypothermia Maintained (N=52) | Randomized to Normothermia and Normothermia Maintained (N=45) | Randomized to Hypothermia and Then Excluded (N=67) | Randomized to Normothermia Then Excluded (N=68)
Elevated Intracranial Pressure (Nervous system disorders) | 23 (244) | 18 (128) | 8 (82) | 7 (30) — Intracranial pressure > 20 mm Hg for 2 or more consecutive hours but that does not meet the definition of critical elevated intracranial pressure (See serious adverse events for that definition)
Decreased Cerebral Perfusion Pressure (Nervous system disorders) | 3 (36) | 3 (20) | 5 (31) | 1 (1) — Cerebral perfusion pressure <60 mm Hg for 2 or more consecutive hours but that does not meet the definition of critical decreased perfusion pressure (See serious adverse events for that definition)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 28 (29) | 28 (33) | 17 (20) | 17 (19) — new or progressive infiltrated, consolidation or pleural effusion on chest x-ray and at least one of the following: 1. New onset of purulent sputum 2. isolation of a etiologic agent 3. Diagnostic antibody titer or detection of viral antigen
Urinary Tract Infection (Renal and urinary disorders) | 3 (5) | 6 (6) | 5 (5) | 4 (4) — Fever >38C and positive urine culture or physician diagnosis of urinary tract infection
Deep Vein Thrombosis (Vascular disorders) | 6 (6) | 6 (6) | 0 (0) | 2 (2) — diagnostic (ultrasound, venogram, Doppler studies) evidence of deep vein thrombosis
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (5) | 0 (0) | 2 (2) — presence of air in the pleural cavity which is not present on admission x-ray and is not associated with hypoxemia or respiratory distress
Decubitus (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2) | 4 (4) | 2 (2) — new ulceration of the skin and subcutaneous tissue which is pressure-related; code only Stage II ulcers or higher (through epidermis and dermis)
hypotension (General disorders) | 7 (8) | 3 (7) | 6 (10) | 4 (21) — Systolic blood pressure <90 mm Hg or Mean arterial pressure <70 mm Hg for 2 or more consecutive hours but not associated with end-organ failure due to hypoperfusion (see Serious Adverse events for definition of critical hypotension)

LIMITATIONS AND CAVEATS:
Early termination for futility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No